CLINICAL TRIAL: NCT04575038
Title: The CRISIS2 Study: A Phase 2, Randomized, Double Blind, Placebo-controlled, Multi-center Study Assessing the Safety and Anti-coronavirus Response of Suppression of Host Nucleotide Synthesis in Out-patient Adults With SARS-CoV-2
Brief Title: CRISIS2: A Phase 2 Study of the Safety and Antiviral Activity of Brequinar in Non-hospitalized Pts With COVID-19
Acronym: CRISIS2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clear Creek Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCB-CRISIS-02
Record Dates: First submitted 2020-10-01; First posted 2020-10-05 (Actual); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — brequinar

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 brequinar 100 mg or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brequinar 100 mg (Experimental): Brequinar oral capsules 100 mg x 5 days
  Interventions: Drug: Brequinar
- Placebo (Placebo Comparator): Placebo for Brequinar capsules x 5 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brequinar — Dihydroorotate dehydrogenase inhibitor (DHODHi)
  Arms: Brequinar 100 mg
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of DHODHi (brequinar) as an antiviral via 5 days of treatment of participants with positive COVID-19 and at least one symptom of COVI019 in an out-patient setting. The study is multi-center, randomized, and placebo-controlled.

DETAILED DESCRIPTION:
Brequinar is a potent DHODH inhibitor that has been previously studied in more than 1,000 cancer, psoriasis, and organ transplant patients. Brequinar has been found to have potent in vitro antiviral activity against many RNA viruses including SARS-CoV-2. The antiviral activity of brequinar against SARS-CoV-2 is likely due to DHODH inhibition and shows nanomolar potency and a high selectivity index in inhibiting viral replication in in vitro studies.

The CRISIS2 trial will study out-patients (non-hospitalized patients) who have a positive SARS-CoV-2 test and are symptomatic. Subjects will be randomized to receive standard of care (SOC) + 5 days of brequinar or SOC + 5 days of placebo. The purpose of this study is to determine if the in vitro antiviral activity of brequinar can be duplicated in patients infected with SARS-CoV-2 by measuring the effect of brequinar on viral shedding. Importantly, the safety and tolerability of brequinar will also be determined in these patients. The results of this proof-of-concept study will inform future studies that will help determine if brequinar is a safe and effective drug for the treatment of SARS-CoV-2 infection.

This will be a phase II randomized, placebo-controlled, double blind, multi-center study with approximately 100 subjects. All subjects will receive standard of care (SOC) per institutional guidelines for treatment of patients with COVID-19 infection. In addition to SOC, the subjects will self-administer one capsule once daily for 5 days.

Subjects will have a Screening Visit followed as soon as possible with Study Day 1. Study visits (virtual or in person) will take place at Screening and on specified days. The visits that include bloodwork must be conducted at the study site or arrangements made for sample collection at the subject's home or other appropriate location. Other visits/visit activities for that visit may be conducted remotely using telemedicine or other remote technique. Subjects are to self-collect a viral load sample, obtain their respiratory rate, heart rate, body temperature and SpO2, and complete a symptom assessment checklist on specified days.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent for the trial, written, electronic, verbal or other method deemed acceptable by the institution and IRB.
2. 18 years of age or older.
3. Laboratory-confirmed SARS-CoV-2 infection as determined by real time polymerase chain reaction (RT-PCR) or other FDA-approved commercial or public health assay.
4. Out-patient (never hospitalized as an in-patient for COVID-19 or was evaluated/treated for COVID-19 only in the Emergency Room with a stay of < 24 hours)
5. The effects of brequinar on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation, and for 90 days after completion of brequinar administration.
6. Male subjects must agree to refrain from sperm donation and female subjects must agree to refrain from ovum donation from initial study drug administration until 90 days after the last dose of brequinar.
7. Must have at least one COVID-19 symptom including but not limited to fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, shortness of breath, dyspnea, anosmia, dysgeusia, or other symptom commonly associated with COVID-19 in the opinion of the investigator. Symptom onset must be ≤7 days prior to first dose. Subject must have one or more symptoms at first dose.
8. Able to swallow capsules.

Exclusion Criteria:

1. Any physical examination findings and/or history of any illness that, in the opinion of the study investigator, might confound the results of the study or pose an additional risk to the patient
2. Nursing women or women of childbearing potential (WOCBP) with a positive pregnancy test
3. Treatment with another DHODH inhibitor (e.g., leflunomide, teriflunomide) or other agents known to cause bone marrow suppression leading to thrombocytopenia
4. Platelets ≤150,000 cell/mm3
5. Hemoglobin < 10 gm/dL
6. Absolute neutrophil count < 1500 cells/mm3
7. Renal dysfunction, i.e., creatinine clearance < 30 mL/min
8. AST or ALT > 2 x ULN, or total bilirubin > ULN. Gilbert's Syndrome is allowed.
9. Bleeding disorders or blood loss requiring transfusion in the six weeks preceding enrollment
10. Ongoing gastrointestinal ulcer, or gastrointestinal bleeding within 6 weeks of randomization.
11. Chronic hepatitis B infection, active hepatitis C infection, active liver disease and/or cirrhosis per subject report.
12. Heart failure, current uncontrolled cardiovascular disease, including unstable angina, uncontrolled arrhythmias, major adverse cardiac event within 6 months (e.g. stroke, myocardial infarction, hospitalization due to heart failure, or revascularization procedure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Central Alabama Research, Homewood, Alabama
  - Ark Clinical Research, Long Beach, California
  - Doral Medical Research, Doral, Florida
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - Monroe Biomedical Research, Monroe, North Carolina
  - Wilmington Health, Wilmington, North Carolina
  - Remington-Davis, Inc., Columbus, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - VitaLink - Gaffney, Gaffney, South Carolina
  - Self Regional Healthcare Research Center - Self Medical Group, Greenwood, South Carolina
  - VitaLink Research, Spartanburg, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Centex Studies, Inc. - McAllen, McAllen, Texas
  - Synexus Clinical Research US, Inc. - Olympus Family Medicine, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were all confirmed to be positive for COVID-19 by means of either a rapid antigen or RT-PCR test. Subjects were out-patients (not hospitalized) at the time of study entry. The first subject was enrolled on 19-NOV-2020; the last subject completed the study on 29-MAR-2021.
Pre-assignment Details: A total of 182 subjects were screened for the study at 14 centers in the US. The Screening period was not more than 7 days in order to provide subjects the earliest possible opportunity for antiviral treatment. The primary screen fail reason was failure to meet one of the laboratory eligibility criteria including low hemoglobin, low platelets, low neutrophil count, and elevated liver function test. Qualifying subjects were enrolled into the study and randomized on the same day.
Groups:
- Standard of Care + Brequinar 100 mg: Standard of Care + Brequinar oral capsules 100 mg x 5 days
  Brequinar: Dihydroorotate dehydrogenase inhibitor (DHODHi)
- Standard of Care + Placebo: Standard of Care + Placebo for Brequinar oral capsules x 5 days
  Placebo: Placebo capsules
Period: Overall Study
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
Started | 56 | 59
Completed | 55 | 58
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Population was used for efficacy analyses. The ITT Set consisted of all randomized subjects. ITT subjects were analyzed according to their randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo | Total
Number analyzed (Participants) | 56 | 59 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 105
  >=65 years | 3 | 7 | 10
Age, Continuous [Median (Full Range); unit: years] | 46.5 [20 to 70] | 45.0 [19 to 83] | 46.0 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 22 | 59
  Male | 19 | 37 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 36
  Not Hispanic or Latino | 38 | 41 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 12 | 14
  White | 53 | 45 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 56 | 59 | 115
Detectable Log 10 SARS-CoV-2 Viral Load [Count of Participants; unit: Participants]
  Detectable | 43 | 45 | 88
  Undetectable | 7 | 12 | 19
  Inconclusive | 0 | 0 | 0
  Missing | 6 | 2 | 8
Body Temperature [Median (Full Range); unit: Degrees Celsius] | 36.7 [34.4 to 37.9] | 36.7 [35.1 to 39.4] | 36.7 [34.4 to 39.4]
SpO2 [Median (Full Range); unit: Percentage of blood oxygen saturation] | 98.0 [93 to 99] | 97.0 [91 to 99] | 98.0 [91 to 99]
Respiratory Rate [Median (Full Range); unit: Breaths per minute] | 16.0 [12 to 30] | 16.0 [10 to 32] | 16.0 [10 to 32]
COVID-19 Symptom Type [Count of Participants; unit: Participants]
  Cough | 43 | 44 | 87
  Headache | 44 | 40 | 84
  Malaise | 44 | 39 | 83
  Sore Throat | 28 | 34 | 62
  Anosmia | 25 | 28 | 53
  Muscle Pain | 23 | 22 | 45
  Gastrointestinal Symptoms | 22 | 21 | 43
  Fever | 18 | 23 | 41
  Shortness of Breath | 19 | 22 | 41
  Dysgeusia | 18 | 17 | 35
  Chills/Rigors | 17 | 15 | 32
  Nasal Congestion | 6 | 10 | 16
  Dyspnea | 5 | 0 | 5
  Fatigue | 5 | 4 | 9
  Body Aches | 0 | 0 | 0
  Other | 12 | 13 | 25
WHO Ordinal Scale [Count of Participants; unit: Participants] — The World Health Organization (WHO) Ordinal Scale provides a high-level categorization of a subject's overall status in terms of:
  Score of 0 = Uninfected; No Viral RNA detected; Score of 1 = Ambulatory Mild Disease - Asymptomatic; Viral RNA detected; Score of 2 = Ambulatory Mild Disease - Symptomatic; Independent; Score of 3 = Ambulatory Mild Disease - Symptomatic; Assistance Needed; Missing
  Participants
    WHO Score of 0 | 0 | 0 | 0
    WHO Score of 1 | 0 | 0 | 0
    WHO Score of 2 | 52 | 52 | 104
    WHO Score of 3 | 0 | 0 | 0
    Missing | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Log10 SARS-CoV-2 Viral Load
Description: Median Change from Baseline in Quantitative Log10 SARS-CoV-2 viral load at Days 4, 8, 12, 15, 22, and 29.
Time Frame: Days 4, 8, 12, 15, 22, and 29
Population: Microbiology Evaluable Set (MES) consisted of all randomized subjects with detectable Log10 SARS-CoV-2 viral load at baseline and at least one non-missing postbaseline viral load assessment. Microbiology evaluable subjects were analyzed according to their randomized treatment. SARS-CoV-2 viral load (log 10 copies/mL) was reported as below.
  * Number of copies/mL;
  * <Number of copies/mL, if detected but under the lower limit of quantification (LLOQ);
  * No SARS-CoV-2 detected, if not detected.
Measure: Median (Full Range); unit: Log 10 SARS-CoV-2 Viral Load Copies/mL
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
Number analyzed (Participants) | 43 | 45
Log 10 SARS-CoV-2 Viral Load Copies/mL
  Baseline | 5.056 [3.14 to 7.96] | 5.110 [3.14 to 8.22]
  Day 4 Change from Baseline: number analyzed (Participants) | 39 | 40
  Day 4 Change from Baseline | -1.651 [-7.94 to 0.87] | -1.881 [-7.21 to 0.93]
  Day 8 Change from Baseline: number analyzed (Participants) | 34 | 38
  Day 8 Change from Baseline | -2.413 [-7.94 to 1.85] | -3.231 [-7.78 to 0.12]
  Day 12 Change from Baseline: number analyzed (Participants) | 37 | 34
  Day 12 Change from Baseline | -3.907 [-7.94 to 0.45] | -3.514 [-7.78 to 0.00]
  Day 15 Change from Baseline: number analyzed (Participants) | 36 | 39
  Day 15 Change from Baseline | -4.140 [-7.94 to 0.20] | -3.143 [-7.78 to 1.40]
  Day 22 Change from Baseline: number analyzed (Participants) | 36 | 41
  Day 22 Change from Baseline | -4.874 [-7.94 to 0.26] | -3.575 [-7.78 to -0.31]
  Day 29 Change from Baseline: number analyzed (Participants) | 38 | 40
  Day 29 Change from Baseline | -4.170 [-7.94 to 3.09] | -3.839 [-7.78 to -1.20]

2. Secondary Outcome: Rates of AEs and SAEs Including Laboratory Assessments
Description: Safety measured by number of participants with AEs and SAEs including laboratory assessments.
Time Frame: Through Day 29
Population: The Safety Analysis Set (Safety) consisted of all subjects who received at least one dose of study drug. Safety analysis subjects were analyzed according to their actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
Number analyzed (Participants) | 56 | 59
Participants
  Any AE | 10 | 13
  Maximum Grade 1 AE | 8 | 8
  Maximum Grade 2 AE | 1 | 2
  Maximum Grade 3 AE | 1 | 3
  Maximum Grade 4 AE | 0 | 0
  Maximum Grade 5 AE | 0 | 0
  Study Drug-Related AE | 3 | 3
  AE Leading to Study Drug Discontinuation | 0 | 0
  Severity Grade 3 or Higher Study Drug Related AE | 0 | 0
  SAE | 1 | 0

3. Secondary Outcome: Viral Shedding Duration
Description: Duration of viral shedding was defined as the time to viral clearance (two consecutive negative test results) for the Microbiology Evaluable Set population.
Time Frame: Through Day 36
Population: Microbiology Evaluable Set (MES) consisted of all randomized subjects with detectable Log10 SARS-CoV-2 viral load at baseline and at least one non-missing postbaseline viral load assessment. Microbiology evaluable subjects were analyzed according to their randomized treatment.
Measure: Median (Full Range); unit: Days
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
Number analyzed (Participants) | 43 | 45
Days | 12.0 [4 to 29] | 8.0 [4 to 36]

4. Secondary Outcome: Hospital Admission
Description: Percentage of subjects requiring admission as an inpatient for >24 hours
Time Frame: Day 29
Population: Intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
Number analyzed (Participants) | 56 | 59
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: 29 Days
Arm/Group | Standard of Care + Brequinar 100 mg | Standard of Care + Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/56 | 0/59
Other Adverse Events (participants affected / at risk) | 3/56 | 4/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care + Brequinar 100 mg (N=56) | Standard of Care + Placebo (N=59)
COVID-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care + Brequinar 100 mg (N=56) | Standard of Care + Placebo (N=59)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04575038/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04575038/SAP_001.pdf